CLINICAL TRIAL: NCT06635811
Title: Circadian Adaptive Deep Brain Stimulation in Essential Tremor
Brief Title: Circadian Adaptive DBS in Essential Tremor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB202400652
Record Dates: First submitted 2024-09-13; First posted 2024-10-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Essential Tremor
Keywords: deep brain stimulation; adaptive DBS
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Adaptive DBS, Then Conventional DBS (Experimental): Participants will initially have their DBS programmed to automatically turn off during sleep for 2 weeks. Then, they will transition to continuous stimulation for another 2 weeks.
  Interventions: Device: Circadian Adaptive DBS; Device: Conventional DBS
- Conventional DBS, then Adaptive DBS (Experimental): Participants will initially have their DBS programmed with continuous stimulation for 2 weeks. Then, they will transition to having their DBS automatically turned off during sleep for another 2 weeks.
  Interventions: Device: Circadian Adaptive DBS; Device: Conventional DBS

INTERVENTIONS:
Device: Circadian Adaptive DBS — DBS automatically turned off during sleep
Device: Conventional DBS — Continous DBS

SUMMARY:
Deep brain stimulation (DBS) of the thalamus is an effective treatment for medically refractory essential tremor (ET). DBS involves delivering continuous stimulation to the brain through electrodes permanently implanted in the thalamus. Despite proven effectiveness, the long-term benefit of DBS can wane over time (habituation) and side effects, including paresthesia and dysarthria, often limit the amplitude of the stimulation, resulting in suboptimal control of tremor. In clinical practice, many groups advise patients to switch their devices off at night to avoid habituation and reduce side effects. However, manually turning off the device at night can result in uncontrolled tremor when the patient moves at night.

This study aims to develop an algorithm that automatically turns off stimulation when a patient is asleep, based on circadian brain signals. Turning off stimulation could potentially improve the therapy by limiting adverse effects, increasing efficacy, reducing the risk of habituation, and prolonging battery life. This study will evaluate the feasibility, safety, and tolerability of circadian adaptive DBS.

DETAILED DESCRIPTION:
This single-center study will investigate the feasibility of developing an adaptive Deep brain stimulation (aDBS) strategy using thalamic circadian rhythm as a control signal. It will evaluate the safety and tolerability of aDBS compared to conventional DBS (cDBS) in a double-blinded cross-over design.

This study will recruit 25 Essential Tremor (ET) patients implanted with the bidirectional neural interface, Medtronic Percept PC (FDA approved), attached to DBS directional lead(s) (Sensight) implanted unilaterally or bilaterally in the ventral intermediate nucleus (VIM) and who are receiving adequate control of their tremor with VIM DBS.

First, the brain signal will be recorded for 1 month to identify circadian fluctuations that may be used to identify the period of sleep. Second, for each patient, an aDBS algorithm based on individualized brain activity will be developed and tested for 2 weeks in a double-blinded cross-over design comparing aDBS and cDBS. Third, at the end of this 4-week trial, patients who preferred aDBS will have the opportunity to stay on aDBS for 6 months, allowing to assess the long-term tolerability of the aDBS.

Each patient enrolled in this study will participate in 7 study visits over 8 months during which chronic brain recordings and aDBS will be set up. Symptoms and stimulation-induced side effects will be assessed by clinicians during these visits. Self-rating scales and wearable will be provided to track tremor, sleep, and movement at home.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Essential Tremor confirmed by a Movement Disorders specialist following established criteria recommended by the Movement Disorders Society
* Patients implanted with unilateral or bilateral VIM DBS leads attached to the Medtronic Percept DBS device for the treatment of Essential Tremor
* Patients with clinical benefit of DBS as defined by a 30% improvement on the TRS or TETRAS at least 3 months after DBS implantation
* DBS programmed in a monopolar configuration allowing chronic brain sensing (C+1- or C+2- in ring mode or any direction)
* Be between 21 and 89 years old
* Ability to give informed consent for the study

Exclusion Criteria:

* Inability to comply with the study protocol
* Pregnancy: all women of childbearing potential will have a negative urine pregnancy test prior to undergoing the study
* Current active suicidal ideation (Yes to #2-5 on C-SSRS)
* Any personality or mood symptoms that study personnel believe will interfere with study requirements

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Presence of thalamic circadian rhythm | Baseline (first month of study participation)
  Thalamic circadian rhythm is defined as a significant difference in day vs night brain activity. It can be used to set up adaptive DBS.
Incidence of stimulation-induced adverse events with aDBS compared to cDBS | Double-blind crossover period (second month of study participation)
  Adverse events are monitored the entire time subject is enrolled in study. Stimulation-induced adverse events during the double-blind crossover is a primary endpoint.

SECONDARY OUTCOMES:
Patient's quality of life as assessed by the Quality of Life in Essential Tremor Questionnaire (QUEST), adapted for a 2-week assessment | From enrollment to the end of study (8 months)
  The QUEST is designed to evaluate the impact of essential tremor on daily functioning and well-being. The total score ranges from 0 to 120, with higher scores indicating worse quality of life.
The Tremor Research Group Essential Tremor Rating Scale (TETRAS) Activities of Daily Living Subscale | From enrollment to the end of study (8 months)
  The TETRAS Activities of Daily Living Subscale will assess the ability to perform daily tasks. The total score ranges from 0 to 48, with higher scores indicating greater difficulty in performing tasks.
Sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI), adapted for a 2-week assessment | From enrollment to the end of study (8 months)
  The PSQI is used to assess the quality of sleep. PSQI score ranges from 0 to 21, with higher scores indicating poorer sleep quality. Each of the seven components of the PSQI is scored from 0 to 3, with 3 indicating the greatest dysfunction.
Patient's cognition as assessed by the Montreal Cognitive Assessment 5-Minute Protocol (Mini MoCA) | From enrollment to the end of study (8 months)
  The Mini MoCA will be used to evaluate cognitive function in patients. It assesses short-term memory, executive function, verbal fluency, attention, and orientation. Scores range from 0 to 30, with higher scores indicating better cognitive performance.
Patient's mood as assessed by the Beck Depression Inventory-II (BDI-II), adapted for a 2-week assessment | From enrollment to the end of study (8 months)
  The BDI-II will be used to assess depressive symptoms in patients. The questionnaire consists of 21 items, each rated on a scale from 0 to 3. Total scores range from 0 to 63, with higher scores indicating more severe depression. Scores are categorized as minimal (0-13), mild (14-19), moderate (20-28), and severe (29-63).
Patient's impression as assessed by the Patient Global Impression of Change Scale (PGI-C) | From enrollment to the end of study (8 months)
  The PGI-C will be used to evaluate the patient's perception of improvement or worsening over time. The PGI-C is rated on a 7-point Likert scale, ranging from 1 (very much improved) to 7 (very much worse). Lower scores indicate better-perceived improvement, while higher scores reflect deterioration.
Patient's self-report of side effects, tremor severity, and sleep | From enrollment to the end of study (8 months)
  At each study visit symptoms are assessed using our Custom Symptom Questionnaire (CSQ). Additionally, during the double-blind crossover period, side effects, tremor severity, and sleep is assessed daily using our Daily Assessment scale.
Presence/severity of tremor tracked with wearable device | From enrollment to the end of double-blind crossover period (first two months of study)
  Subjects will be given a wearable device, a Fitbit watch, for objective assessment of tremor.
Battery drainage/Stimulation energy use as assessed by Total Electrical Energy Delivered (TEED) | From enrollment to the end of study (8 months)
  The TEED will be calculated and compared for both aDBS and cDBS over a 2-week period. TEED is measured in millijoules (mJ), and lower values indicate lower energy consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Norman Fixel Institute for Neurological Diseases, Gainesville, Florida, United States